CLINICAL TRIAL: NCT02010307
Title: Polymorphonuclear Cells' Sensitivity to Aggregatibacter Actinomycetemcomitans Bacteria in Patients With Aggressive Periodontitis
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Polak David (Other)
Responsible Party: Sponsor-Investigator, Polak David, senior dentist, periodontology department, Hadassah Medical Organization
Organization: Hadassah Medical Organization (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: davidp-HMO-CTIL
Record Dates: First submitted 2013-12-09; First posted 2013-12-12 (Estimated); Last update posted 2013-12-16 (Estimated); Status verified 2013-12

CONDITIONS: Periodontal Disease
MeSH Terms: conditions — Periodontal Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- aggressive periodontitis (Experimental): 25 patients with aggressive periodontitis blood extraction
  Interventions: Other: blood extraction
- chronic periodontitis (Experimental): 25 patients with chronic periodontitis blood extraction
  Interventions: Other: blood extraction
- healthy (Experimental): 25 healthy periodontal patients blood extraction
  Interventions: Other: blood extraction

INTERVENTIONS:
Other: blood extraction — 6 ml blood extraction from each patients in all 3 arms of the study

SUMMARY:
aggressive periodontitis is an inflammatory disease which damage the teeth supporting structures mostly in young patients. and has genetic basis.

a specific bacteria: Aggregatibacter actinomycetemcomitans (Aa) is associated with this disease, and found to damage leukocytes by using a specific leukotoxin.

in the research the investigators are aiming to find molecular and immunological basis to aggressive periodontitis.

ELIGIBILITY:
Inclusion Criteria:

* patients in periodontal department
* healthy
* diagnosed with chronic/aggressive periodontal disease
* interested in participating the research

Exclusion Criteria:

* diagnosed with diabetes, heart disease, immunosuppression, thrombocytopenia, clotting enzyme deficiency.
* using alcohol, or drugs
* pregnancy

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 75 (Estimated)
Dates: Start 2014-01; Primary Completion 2015-01 (Estimated); Study Completion 2015-10 (Estimated)

PRIMARY OUTCOMES:
flow cytometry | 12 hours after blood extraction
  the investigators use flow cytometry technique in order to determine the influence of gingival bacteria on the leukocytes, after culturing the two together.

SECONDARY OUTCOMES:
microscopy observation | 12 hours after blood extraction
  the investigators use microscopy in order to determine the influence of gingival bacteria on the leukocytes, after culturing the two together

CONTACTS AND LOCATIONS:
Overall Officials: David Polak, DMD, PhD, Principal Investigator — Haddasah Medical Center
Locations (1):
- Hadassah Medical Organization, Jerusalem, Israel, Jerusalem, Israel